CLINICAL TRIAL: NCT06340425
Title: The Effect of Selective Dorsal Rhizotomy on a Multidimensional Outcome Set in Children With Spastic Cerebral Palsy: a Retrospective Study
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Kaat Desloovere, prof. dr., Universitaire Ziekenhuizen KU Leuven
Other Study IDs: s68727
Record Dates: First submitted 2024-03-01; First posted 2024-04-01 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Cerebral Palsy
Keywords: Cerebral palsy; Selective dorsal rhizotomy; Spasticity; Muscle morphology; Gait; Gross motor function; Clinical examination
MeSH Terms: conditions — Cerebral Palsy; Muscle Spasticity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SDR group, main group will be evaluated within subject design: * Patient characteristics: Children with spastic cerebral palsy, 5 to 16 years of age at time of SDR, both male and female. All children were diagnosed with bilateral involvement, Gross Motor Function Classification System level II or III.
  * Intervention: All participants underwent an SDR procedure in terms of their clinical care, based on the clinical decision making of the attending physician. During the SDR procedure, 25-30% of the dorsal rootlets was cut, descending between L1 and S1. Children received an intensive one-year rehabilitation program after the procedure, of which two to three months of the rehabilitation was performed while the child was admitted to the hospital.
  The effects within the SDR group will be compared to two control groups (see below).
- Control groups: Additionally two reference databases, established during previous research, will be used to improve interpretation. A normative reference database of typically developing children will be used to calculate the three-dimensional gait analysis outcomes. This database consists of 87 typically developing children (aged between 4,5 and 18,5 years, 42 boys and 45 girls, weight range 17,6 and 92,5 kg, height range between 1,08 and 1,9 meter). A reference database of children with spastic CP without a SDR intervention will be used to qualitatively judge the muscle morphology of children with spastic CP with an SDR intervention. This database consists of 206 children with CP (aged between 0,6 and 17,4 years, 124 boys and 82 girls, weight range 5,8 and 82,0 kg, height range between 0,6 and 1,9 meter, 88 with unilateral and 118 with bilateral involvement, 104 with a GMFCS level 1, 63 with a level 2 and 39 with a level 3).

SUMMARY:
Cerebral palsy or CP is the single largest cause of childhood physical disability, with a prevalence of 2-3 per 1000 livebirths. Children with CP experience different primary symptoms, including abnormal increased muscle tone or spasticity. Selective dorsal rhizotomy (SDR) is applied in children with spastic CP as a non-reversible tone reduction procedure. Better understanding of the effects of SDR on a multidimensional outcome set in one CP-cohort and on macroscopic muscle morphology can improve insights and clinical decision making.

DETAILED DESCRIPTION:
Cerebral palsy or CP is the single largest cause of childhood physical disability, with a prevalence of 2-3 per 1000 livebirths. Children with CP experience different primary symptoms, including abnormal increased muscle tone or spasticity. Selective dorsal rhizotomy (SDR) is applied in children with spastic CP as a non-reversible tone reduction procedure. During this neurosurgical procedure, dorsal rootlets are transected to diminish the excitatory input from the afferents, resulting in a reduction of the abnormal, increased muscle tone. Although different studies investigated the SDR-effect on separate sets of outcomes, such as spasticity, gait or gross motor function, no study so far has studied SDR-effects on combined outcome sets in one CP-cohort or on macroscopic muscle morphology.

The discrepancy between results of different previous studies highlight the added value of a multidimensional outcome set assessed within one cohort. Integrating outcomes of different levels will provide a better insight on how effects do or do not occur. Additionally, although SDR does not directly intervene with the macroscopic muscle structures, reducing the excitatory input from the afferents could potentially have an effect on muscle growth. Indicating macroscopic muscle morphology as an important outcome.

The current study will investigate the added value of a multidimensional outcome set, assessed in one single cohort. Important gaps in the literature will be addressed, including the effect of SDR on muscle morphology and the use of instrumented assessments. The primary objective of this study was to investigate changes in a multidimensional outcome set (including spasticity, muscle morphology, gait and gross motor function) pre- and post-SDR, in one single cohort of children with spastic CP. As a secondary objective, this study will compare outcomes of the clinical examination (spasticity, range of motion, strength, selectivity) pre- and post-SDR. Additionally, muscle morphology will be qualitatively compared in children with CP who received an SDR to children with CP without an SDR intervention.

ELIGIBILITY:
Inclusion Criteria:

* Spastic CP, Uni- or bilateral involvement
* Gross Motor Classification System (GMFCS) levels I to III
* Children: 5 to 16 years of age at time of SDR
* SDR intervention
* Clinical follow-up pre- and post-SDR at the Clinical Motion Analysis Laboratory Pellenberg (CMAL, UZ Leuven, Campus Pellenberg)

Exclusion Criteria:

* Presence of dystonia or ataxia
* SDR intervention in combination with muscle surgery
* Severe co-morbidities (that are likely to prevent proper assessment, such as severe cognitive problems)

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with spastic cerebral palsy, receiving SDR at the CP reference center of the University Hospitals Leuven and have clinical follow-up pre- and post-SDR at the Clinical Motion Analysis Laboratory Pellenberg (CMAL, UZ Leuven, Campus Pellenberg)
  Control groups:
  * Reference database of children with spastic cerebral palsy, without a SDR intervention
  * Reference database of typically developing children
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2018-06-26 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Overall changes in spasticity | pre- and one year post-SDR
  The specific outcome is the difference in the root mean square value of the surface-EMG signals between the low- and high-velocity passive stretches, expressed both absolute and normalized to the maximum voluntary contraction.
Overall change in muscle volume of the medial gastrocnemius | pre- and one year post-SDR
  Estimation of the muscle belly volume, measured by 3DfUS. Muscle volume will be expressed absolute and normalized to anthropometric growth.
Overall changes in muscle length of the medial gastrocnemius | pre- and one year post-SDR
  Estimation of the muscle belly length, tendon length and muscle tendon unit complex length, measured by 3DfUS. Muscle lengths will be expressed absolute and normalized to anthropometric growth.
Overall changes in muscle cross-sectional area at 50% of muscle belly length | pre- and one year post-SDR
  Estimation of the muscle belly cross-sectional area at 50% of the muscle belly length, measured by 3DfUS. Muscle cross-sectional area will be expressed absolute and normalized to anthropometric growth.
Overall changes in gait | pre- and one year post-SDR
  Gait was measured with three-dimensional gait analysis. The specific outcomes are the gait profile score and the gait variable scores of the ankle and the knee. Parameters were calculated using the reference database of typically developing children.
Overall change in gross-motor function | pre- and one year post-SDR
  Gross-motor function was measured with the Gross-motor function measure 66- item set, resulting in a total score.

SECONDARY OUTCOMES:
Overall change of spasticity in the plantar flexors | pre- and one year post-SDR
  Evaluation of spasticity of the plantar flexors, measured with the Modified Ashworth Scale.
Overall change of selectivity in the plantar flexors | pre- and one year post-SDR
  Evaluation of selectivity of the plantar flexors, measured with the selective motor control test.
Overall change of passive range of motion in the ankle and knee joint | pre- and one year post-SDR
  Evaluation of passive range of motion in the ankle and knee joint, measured by goniometry.
Overall change of muscle strength in the plantar flexors | pre- and one year post-SDR
  Evaluation of muscle strength of the plantar flexors, measured with the Medical Research Council Scale.
Scatter plots of muscle morphology data (same parameters as for the primary endpoints) | SDR (pre- and one year post-SDR )vs no SDR (a database of children with CP who were not treated with SDR, one timepoint)
  Scatter plots of muscle morphology data per age, for the reference database of children with spastic cerebral palsy, without an SDR intervention, overlaid by the individual data points of the enrolled children with CP who did receive an SDR intervention, pre and 1 year post SDR.

CONTACTS AND LOCATIONS:
Overall Officials: Kaat Desloovere, prof. dr., Principal Investigator — Department of Rehabilitation Sciences, KU Leuven, Belgium
Locations (1):
- UZ Leuven, Leuven, Vlaams-Brabant, Belgium